CLINICAL TRIAL: NCT01797081
Title: BOTOX® in the Treatment of Crow's Feet Lines in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-114
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Lateral Canthus Rhytides; Crow's Feet Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Botulinum toxin Type A (24U) (Experimental): 24 units (U) botulinum toxin Type A (total dose) injected into bilateral Crow's Feet Line areas on Day 1. Based on retreatment criteria participants were eligible for up to 5 treatment cycles.
  Interventions: Biological: botulinum toxin Type A (24 U)
- Botulinum toxin Type A (12U) (Experimental): 12U botulinum toxin Type A (total dose) injected into bilateral Crow's Feet Line areas on Day 1. Based on retreatment criteria participants were eligible for up to 5 treatment cycles.
  Interventions: Biological: botulinum toxin Type A (12 U)
- Placebo/Botulinum toxin Type A (24U) (Other): Placebo (normal saline) one treatment injected into bilateral Crow's Feet Line areas on Day 1 and subsequent treatments if applicable until day 180. Botulinum toxin Type A (24U) injected into bilateral Crow's Feet Line areas at any additional treatments from day 180 onward. Based on retreatment criteria participants were eligible for up to 5 treatment cycles (2 Placebo + 3 botulinum toxin type A).
  Interventions: Biological: botulinum toxin Type A (24 U); Other: Normal Saline
- Placebo/Botulinum toxin Type A (12U) (Other): Placebo (normal saline) one treatment injected into bilateral Crow's Feet Line areas on Day 1 and subsequent treatments if applicable until day 180. Botulinum toxin Type A (12U) injected into bilateral Crow's Feet Line areas at any additional treatments from day 180 onward. Based on retreatment criteria participants were eligible for up to 5 treatment cycles (2 Placebo + 3 botulinum toxin type A).
  Interventions: Biological: botulinum toxin Type A (12 U); Other: Normal Saline

INTERVENTIONS:
Biological: botulinum toxin Type A (24 U) — 24 units botulinum toxin Type A (total dose) injected into bilateral Crow's Feet Line areas per treatment.
  Other Names: BOTOX®
  Arms: Botulinum toxin Type A (24U); Placebo/Botulinum toxin Type A (24U)
Biological: botulinum toxin Type A (12 U) — 12 units botulinum toxin Type A (total dose) injected into bilateral Crow's Feet Line areas per treatment.
  Other Names: BOTOX®
  Arms: Botulinum toxin Type A (12U); Placebo/Botulinum toxin Type A (12U)
Other: Normal Saline — Normal saline (placebo) injected into bilateral Crow's Feet Line areas per treatment.
  Arms: Placebo/Botulinum toxin Type A (12U); Placebo/Botulinum toxin Type A (24U)

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® (botulinum toxin Type A) compared to placebo for the treatment of Crow's Feet Lines (Lateral Canthus Rhytides).

ELIGIBILITY:
Inclusion Criteria:

-Moderate to severe Crow's Feet Lines

Exclusion Criteria:

* Current or previous botulinum toxin treatment of any serotype
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis
* Facial laser or light treatment for cosmetic purposes, microdermabrasion, superficial peels, or topical retinoid therapy or hormone cream within 3 months
* Laser treatment or phototherapy of the face for medical purposes, blepharoplasty, brow-lift or related procedure, periorbital permanent make-up, or oral retinoid therapy within one year
* Medium-depth or deep facial peels within 5 years
* Prior facial cosmetic surgery (e.g., prior periorbital surgery, facial lift, periorbital treatment with fillers, implantation or transplantation)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2013-07-18 (Actual); Study Completion 2014-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Background] Harii K, Kawashima M, Furuyama N, Lei X, Hopfinger R, Lee E. OnabotulinumtoxinA (Botox) in the Treatment of Crow's Feet Lines in Japanese Subjects. Aesthetic Plast Surg. 2017 Oct;41(5):1186-1197. doi: 10.1007/s00266-017-0844-9. Epub 2017 Jul 21. PMID 28733805

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Botulinum Toxin Type A (24 U): Placebo (normal saline) one treatment injected into bilateral Crow's Feet Line areas on Day 1 and subsequent treatments if applicable until day 180. Botulinum toxin Type A (24 U) injected into bilateral Crow's Feet Line areas at any additional treatments from day 180 onward. Based on retreatment criteria participants were eligible for up to 5 treatment cycles (2 Placebo + 3 botulinum toxin type A).
- Placebo/Botulinum Toxin Type A (12 U): Placebo (normal saline) one treatment injected into bilateral Crow's Feet Line areas on Day 1 and subsequent treatments if applicable until day 180. Botulinum toxin Type A (12 U) injected into bilateral Crow's Feet Line areas at any additional treatments from day 180 onward. Based on retreatment criteria participants were eligible for up to 5 treatment cycles (2 Placebo + 3 botulinum toxin type A).
Period: Overall Study
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo/Botulinum Toxin Type A (24 U) | Placebo/Botulinum Toxin Type A (12 U)
Started | 104 | 99 | 48 | 49
Completed | 90 | 95 | 43 | 40
Not Completed | 14 | 4 | 5 | 9
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Personal Reasons | 12 | 4 | 4 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo/Botulinum Toxin Type A (24 U) | Placebo/Botulinum Toxin Type A (12 U) | Total
Number analyzed (Participants) | 104 | 99 | 48 | 49 | 300
Age, Customized [Number; unit: participants]
  ≤ 50 years | 53 | 58 | 28 | 30 | 169
  > 50 years | 51 | 41 | 20 | 19 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 70 | 36 | 34 | 224
  Male | 20 | 29 | 12 | 15 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving None or Mild on the Investigator's Assessment of the Severity of Crow's Feet Lines (CFL) at Maximum Smile Using the Facial Wrinkle Scale-Asian (FWS-A)
Description: The Investigator assessed the severity of the patient's Crow's Feet lines at maximum smile using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30 is reported.
Time Frame: Day 30
Population: Intent-to-treat population included all enrolled participants.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo (normal saline) one treatment injected into bilateral Crow's Feet Line areas on Day 1 and subsequent treatments if applicable until day 180.
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo
Number analyzed (Participants) | 104 | 99 | 97
percentage of participants | 68.3 | 56.6 | 8.2

2. Secondary Outcome: Percentage of Participants Achieving a ≥1-Grade Improvement From Baseline on the Investigator's Assessment of the Severity of CFL at Rest Using the FWS-A
Description: The Investigator assessed the severity of the participant's Crow's Feet Lines at rest using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a ≥1-grade improvement from Baseline at Day 30 is reported.
Time Frame: Day 30
Population: Participants from the Intent-to-treat population, all enrolled participants, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo
Number analyzed (Participants) | 99 | 94 | 81
percentage of participants | 61.6 | 43.6 | 17.3

3. Secondary Outcome: Percentage of Participants Much Improved or Very Much Improved in the Subject's Assessment of Appearance of CFL as Measured by the Global Assessment of Change in Crow's Feet Lines
Description: Participants rated the change in their Crow's Feet Lines using the Subject's Global Assessment of Change in Crow's Feet Lines (SGA-CFL) 7-point scale where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse or 7=very much worse. The percentage of participants who reported Much Improved or Very Much Improved at Day 30 is reported.
Time Frame: Day 30
Population: Intent-to-treat population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo
Number analyzed (Participants) | 104 | 99 | 97
percentage of participants | 49.0 | 39.4 | 1.0

4. Secondary Outcome: Percentage of Participants Who Rate Themselves in a Younger Self-Perception of Age Category Than at Baseline
Description: Participants were considered to judge themselves as looking younger if the category change was from "look my current age" at Baseline to "look younger" at Day 30 or from "look older" at Baseline to "look my current age/younger" at Day 30.
Time Frame: Day 30
Population: Intent-to-treat population included all enrolled participants. Only those participants who rated themselves as looking their current age or older at Baseline were included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo
Number analyzed (Participants) | 100 | 95 | 92
percentage of participants | 32.0 | 30.5 | 7.6

ADVERSE EVENTS:
Description: Adverse events that occurred during the BOTOX cycles of the placebo/BOTOX 24U and placebo/BOTOX 12U participants are included in the corresponding BOTOX groups.
Arm/Group | Botulinum Toxin Type A (24U) | Botulinum Toxin Type A (12U) | Placebo
Serious Adverse Events (participants affected / at risk) | 3/151 | 2/143 | 2/97
Other Adverse Events (participants affected / at risk) | 23/151 | 39/143 | 5/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (24U) (N=151) | Botulinum Toxin Type A (12U) (N=143) | Placebo (N=97)
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (24U) (N=151) | Botulinum Toxin Type A (12U) (N=143) | Placebo (N=97)
Nasopharyngitis (Infections and infestations) | 23 | 39 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.